CLINICAL TRIAL: NCT07082972
Title: Evaluation of the Effects of Occlusal Splint and Masseter Botulinum Toxin Injections on Head and Neck Muscles Using Electromyography
Brief Title: EMG-Based Evaluation of Occlusal Splint and Masseter Botox Effects on Head and Neck Muscles
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Berk Bilgen, Phd DDS, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/150 Rev-1
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Myofascial Pain Syndrome (MPS); Masticatory Muscle Pain
Keywords: Myofascial Pain Syndrome (MPS); Botulinum Toxin; Occlusal Splint; Bruxism; Head and neck muscles; Sternocleidomastoid muscle (SCM); Masseter muscle; Splenius capitis muscle; Electromyography
MeSH Terms: conditions — Myofascial Pain Syndromes; Bruxism | interventions — Botulinum Toxins; Occlusal Splints

STUDY DESIGN:
Intervention Model Description: Patients with myofascial pain syndrome will be included, and their muscle activity will be measured using electromyography (EMG).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Botulinum toxin injection group (Experimental): Patients will receive a total of 20 units of botulinum toxin injected into the masseter muscle on each side. EMG measurements will be taken before and after treatment to evaluate changes in muscle activity.
  Interventions: Drug: Botulinum toxin injection
- Occlusal splint group (Experimental): Patients will use occlusal splints during sleep. EMG recordings will assess the effect of splint therapy on muscle activity.
  Interventions: Device: Occlusal splint
- Botulinum toxin + Occlusal splint combined group (Experimental): Patients will receive 20 units of botulinum toxin injections into the masseter muscle on each side and use occlusal splints during sleep. EMG will monitor the combined effect on muscle activity.
  Interventions: Combination Product: Botulinum toxin + Occlusal splint combined
- Control group (No Intervention): Patients will not receive any active treatment. EMG measurements will observe natural changes over time.

INTERVENTIONS:
Drug: Botulinum toxin injection — Patients will receive a total of 20 units of botulinum toxin type A (Botox) injected into each masseter muscle. The injections will be administered at three standardized sites on each side using a fine needle to ensure accurate delivery. Muscle activity will be recorded using electromyography (EMG) before the injection, and follow-up EMG measurements will be taken at one month and four months post-treatment to evaluate changes in muscle activity and treatment efficacy.
  Arms: Botulinum toxin injection group
Device: Occlusal splint — Patients with myofascial pain syndrome will receive custom-made occlusal splints to wear during sleep. These splints help reduce abnormal muscle activity and relieve pain by redistributing bite forces. EMG measurements will be taken before and during treatment to monitor changes in muscle activity.
  Arms: Occlusal splint group
Combination Product: Botulinum toxin + Occlusal splint combined — Patients will receive both botulinum toxin injections (20 units per masseter muscle, injected at three standardized points per side) and will use occlusal splints during sleep. EMG measurements will be conducted before treatment, and at follow-up visits to assess the combined effect of pharmacological and mechanical therapy on muscle activity.
  Arms: Botulinum toxin + Occlusal splint combined group

SUMMARY:
This randomized controlled clinical trial aims to evaluate the individual and combined effects of occlusal splint therapy and botulinum toxin type A (BTX-A) injections into the masseter muscle on the activity of head and neck muscles in patients diagnosed with myofascial pain syndrome (MPS). MPS is a common subtype of temporomandibular disorders (TMD), frequently involving the masticatory and cervical muscles. Despite various treatment modalities, there is still no universally accepted protocol. In this study, 56 adult participants of both sexes, without missing teeth and within a normal body mass index (BMI) range, will be randomly assigned to four groups: BTX-A injection only, occlusal splint only, combined BTX-A and splint therapy, and an untreated control group. Surface electromyography (EMG) will be used to assess muscle activity in the masseter, temporalis, sternocleidomastoid, splenius capitis, and trapezius muscles. EMG recordings will be performed at baseline, 4 weeks, and 12 weeks after the intervention. Pain levels and symptom severity will be assessed using the DC/TMD symptom questionnaire and the Visual Analog Scale (VAS). BTX-A injections will be administered by a neurology specialist (20 IU per masseter muscle), and occlusal splints will be custom-fabricated and fitted for each participant. This study seeks to determine the neuromuscular effects of these treatments-both alone and in combination-on masticatory and cervical muscles and to provide insight into the development of more comprehensive and effective treatment strategies for MPS.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled, parallel-group clinical trial designed to investigate the effects of occlusal splints and BTX-A injections in adult patients with myofascial pain syndrome (MPS), as diagnosed by the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD). A total of 56 adult participants (both male and female) will be recruited and randomly divided into four equal groups (n=14): (1) BTX-A injection only, (2) occlusal splint only, (3) BTX-A combined with occlusal splint, and (4) control group receiving no treatment. All participants must be within the normal BMI range and have complete dentition.

Exclusion criteria include pregnancy or lactation, systemic neuromuscular or bleeding disorders, prior BTX-A treatment in the masseter region, recent facial aesthetic procedures, and any condition that may hinder study compliance.

BTX-A will be injected into the masseter muscles at three standardized sites per side (total 20 IU per muscle) using a 1 ml syringe with a 26-gauge, 13 mm needle. The injections will be performed by a neurologist in a hospital setting. For participants in the occlusal splint group, upper jaw impressions will be taken using alginate, and splints will be fabricated from 2 mm thick hard vinyl acetate sheets. Splints will be positioned intraorally with autopolymerizing acrylic resin to ensure consistent fit and occlusal contact.

EMG measurements will be conducted at Bezmialem Vakıf University using surface electrodes placed over the masseter, temporalis, sternocleidomastoid, splenius capitis, and trapezius muscles. The skin will be cleaned with 70% alcohol, and electrode placement will follow anatomical landmarks. Recordings will be obtained during maximal voluntary clenching with participants seated and relaxed. Measurements will be taken before treatment, at 4 weeks, and at 12 weeks post-intervention to monitor short- and long-term effects.

All patients will complete the DC/TMD symptom questionnaire and rate their pain using a Visual Analog Scale (VAS) at each time point. Statistical analysis will be performed using SPSS v22. Parametric and non-parametric methods will be applied based on data distribution. Intergroup comparisons will be performed using one-way ANOVA or Kruskal-Wallis tests, and intragroup comparisons will utilize repeated measures ANOVA or Friedman tests. Chi-square tests will be used for categorical data. A significance level of p<0.05 will be considered statistically meaningful.

The study was approved by the Clinical Research Ethics Committee of Istanbul University Faculty of Dentistry and will be funded by the university (BAP). All procedures will be carried out under professional supervision to ensure safety and reliability of data collection.

ELIGIBILITY:
Inclusion Criteria:

1. Having a diagnosis of myofascial pain syndrome
2. No missing teeth
3. No history of previous temporomandibular disorder treatment
4. Absence of an arthrogenic temporomandibular disorder

Exclusion Criteria:

* Pregnancy or lactation; osteoporosis and bisphosphonate use
* Previous botulinum toxin injection to the masseter region
* Bleeding disorders or use of anticoagulant medications
* Presence of systemic muscular or neurological diseases (e.g., myasthenia gravis, ALS)
* Active infection, open wound, or dermatological condition in the facial area
* Undergoing other facial aesthetic procedures (e.g., fillers, PRP, etc.) within the last six months
* Individuals with severe psychiatric disorders or those on regular psychiatric medications
* Patients who are unlikely to comply with the study protocol or complete the follow-up period
* Individuals with a body mass index (BMI) outside the normal range, including underweight or overweight participants, will be excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Electromyography results | 12 week
  Electromyographic (EMG) recordings will be used to assess changes in electrical activity in the masseter, temporalis, sternocleidomastoid (SCM), trapezius, and splenius capitis muscles. These muscles are often overactive in individuals with bruxism, parafunctional habits, and postural issues.
  Baseline EMG recordings will be taken at week 0, with follow-up measurements at the 1st and 12th weeks to observe short- and mid-term effects. EMG activity in the masseter and temporalis muscles will be evaluated to assess changes following botulinum toxin injections, focusing on potential reductions in muscle hyperactivity. Occlusal splint therapy will be analyzed in terms of its effect on normalizing muscle activity over time. The combined treatment group will be examined for additive or prolonged effects. The control group will serve as a reference to monitor natural variations in EMG activity.

SECONDARY OUTCOMES:
Diagnostic Criteria for Temporomandibular Disorders - Clinical Examination Form | 12 week
  Using the DC/TMD Clinical Examination Form, secondary outcomes will be assessed, including the precise location of pain reported by the patients, the characteristics and range of jaw opening movements, as well as the presence and intensity of pain elicited during manual palpation of the masticatory muscles and temporomandibular joint. These evaluations will help to comprehensively understand the functional limitations and pain patterns associated with temporomandibular disorders and will complement the primary outcomes measured in the study.
Evaluation of Pain and Jaw Function as Secondary Outcomes | 12 week
  As another secondary outcome, pain intensity and jaw functional limitations will be evaluated using a validated pain and jaw function limitation questionnaire. This self-reported tool will allow for the assessment of patients' perceived levels of orofacial pain and the impact of temporomandibular disorders on daily jaw functions such as chewing, speaking, and yawning. These data will support the clinical findings and contribute to a more comprehensive understanding of the functional burden caused by myofascial pain.

CONTACTS AND LOCATIONS:
Overall Officials: Olcay Şakar, Phd Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Vezneciler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi KH, Kwon OS, Kim L, Lee SM, Jerng UM, Jung J. Electromyographic changes in masseter and sternocleidomastoid muscles can be applied to diagnose of temporomandibular disorders: An observational study. Integr Med Res. 2021 Dec;10(4):100732. doi: 10.1016/j.imr.2021.100732. Epub 2021 May 16. PMID 34141576
- [Background] Kaya DI, Ataoglu H. Botulinum toxin treatment of temporomandibular joint pain in patients with bruxism: A prospective and randomized clinical study. Niger J Clin Pract. 2021 Mar;24(3):412-417. doi: 10.4103/njcp.njcp_251_20. PMID 33723117
- [Background] Yurttutan ME, Tutunculer Sancak K, Tuzuner AM. Which Treatment Is Effective for Bruxism: Occlusal Splints or Botulinum Toxin? J Oral Maxillofac Surg. 2019 Dec;77(12):2431-2438. doi: 10.1016/j.joms.2019.06.005. Epub 2019 Jun 19. PMID 31302066